CLINICAL TRIAL: NCT00833885
Title: Tolerability and Measurability of the Efficacy of Non Pharmaceutical Measures to Prevent Seasonal Influenza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Koch Institut (Other Government)
Responsible Party: Dr. med. Udo Buchholz, MPH, Robert Koch Institut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RKI-NPI
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Influenza
Keywords: Non pharmaceutical measures
MeSH Terms: conditions — Influenza, Human | interventions — Masks; Hand Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Control
  Interventions: Other: Control
- 2 (Other): Masks
  Interventions: Device: Masks
- 3 (Other): Masks and Hygiene
  Interventions: Device: Masks & hand hygiene

INTERVENTIONS:
Device: Masks — Wearing of surgical masks
  Arms: 2
Device: Masks & hand hygiene — Wearing of surgical masks and intensified hand washing
  Arms: 3
Other: Control — General information about virus transmission in households and basic means to prevent it
  Arms: 1

SUMMARY:
With this study the investigators will try to assess the tolerability and measurability of the efficacy of non pharmaceutical measures to prevent seasonal influenza in individual households. Households with an identified index case of influenza will be randomised into one of three intervention arms: 1. group, where the household will receive general information about transmission of influenza virus and means to prevent it (Controls); 2. group, which will receive surgical masks and be asked to wear them whenever they are in close contact with the index case or other persons of the household that became ill during the observation period; 3. group, which will be given and asked to wear surgical masks as well as to execute intensified hand hygiene.

In addition to assessing the secondary attack rate as our primary outcome measure, the investigators will also try to evaluate compliance to those interventions by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* influenza like illness symptoms
* positive rapid test for influenza
* inclusion within 48h of symptom onset
* inclusion of at least 3 members of a household (including index case)

Exclusion Criteria:

* severe illness
* other cases of similar symptoms within 14 days before onset of symptoms in index patient
* severe asthma or COPD
* pregnancy of index

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Secondary infection with influenza of the household members who are healthy at the start of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Koch Institute, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Jefferson T, Dooley L, Ferroni E, Al-Ansary LA, van Driel ML, Bawazeer GA, Jones MA, Hoffmann TC, Clark J, Beller EM, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2023 Jan 30;1(1):CD006207. doi: 10.1002/14651858.CD006207.pub6. PMID 36715243
- [Derived] Jefferson T, Del Mar CB, Dooley L, Ferroni E, Al-Ansary LA, Bawazeer GA, van Driel ML, Jones MA, Thorning S, Beller EM, Clark J, Hoffmann TC, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2020 Nov 20;11(11):CD006207. doi: 10.1002/14651858.CD006207.pub5. PMID 33215698
- [Derived] Suess T, Remschmidt C, Schink SB, Schweiger B, Nitsche A, Schroeder K, Doellinger J, Milde J, Haas W, Koehler I, Krause G, Buchholz U. The role of facemasks and hand hygiene in the prevention of influenza transmission in households: results from a cluster randomised trial; Berlin, Germany, 2009-2011. BMC Infect Dis. 2012 Jan 26;12:26. doi: 10.1186/1471-2334-12-26. PMID 22280120